CLINICAL TRIAL: NCT05268471
Title: Cost-effectiveness Analysis and Conditional Response to the Effect of Active Postural Devices in Postural Obstructive Sleep Apnea. Pávlov Project.
Brief Title: Cost-effectiveness Analysis and Conditional Response to the Effect of Positional Devices in Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Irene Cano-Pumarega, Sleep Unit Coordinator, Principal Investigator, Clinical Professor, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAVLOV
Record Dates: First submitted 2022-02-08; First posted 2022-03-07 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Positional Device (PD) (Experimental): Vibrating positional device (Nightbalance, Philips) to treat positional obstructive sleep apnea
  Interventions: Device: Positional device (PD)
- Continuos Positive Airway Pressure (CPAP) (Active Comparator): Continuos Positive Airway Pressure (standard treatment) to treat obstructive sleep apnea
  Interventions: Device: Continuos Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Positional device (PD) — OSA treatment with PD for 6 months
  Arms: Positional Device (PD)
Device: Continuos Positive Airway Pressure (CPAP) — OSA treatment with CPAP for 6 months
  Arms: Continuos Positive Airway Pressure (CPAP)

SUMMARY:
The objectives of this study are:

* To assess the effectiveness and cost-effectiveness of a vibrating positional device (NightBalance, Philips) in the treatment of positional obstructive sleep apnea compared to conventional CPAP treatment.
* To investigate whether a positional device (NightBalance, Philips) avoids supine position after a period of use of the device without actively using the device for a subsequent period of time.

DETAILED DESCRIPTION:
Non-inferiority clinical trial open to patients and investigators, multicenter, randomized and controlled to treatment with positional device (PD) and CPAP to evaluate the effectiveness of treatment of positional obstructive sleep apnea with a PD (NightBalance, Philips) compared to CPAP after 6 months of continuous treatment (first phase) and the permanence of such efficacy after subsequent discontinuation of treatment (second phase).

An initial respiratory polygraphy will be performed in all patients and the sleep study will be repeated at 6 months with PD and CPAP. After its withdrawal, in those patients who respond, the respiratory polygraphy will be repeated at one week and one month.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Signed informed consent.
* Diagnosis of POSA by respiratory polygraphy with the following criteria:

  * AHI ≥ 15/h or AHI ≥ 10/h and AHI <15/h with an Epworth >10
  * AHI ns <10/h (<5/h in mild OSA).
  * AHI is at least twice the AHI in ns
  * Time in supine >20%.
  * Valid recording time>4h

Exclusion Criteria:

* Treatment of OSA with CPAP or DAM in the previous month or treatment with surgery for OSA at any time.
* Presence of other sleep disorders or central sleep apnea (central AHI >50% of total AHI).
* Severe cardiovascular, neuromuscular or pulmonary pathology or chronic home oxygen use.
* Poorly controlled arterial hypertension or refractory arterial hypertension.
* Condition that makes it difficult or impossible to change position during sleep.
* Epworth scale score ≥ 16.
* Professional driver, heavy machinery operator or shift worker.
* Pregnancy.
* Treatment with medication that may interfere with alertness or drowsiness such as: sedative antidepressants, hypnotics, opioids, anticonvulsants or central nervous system stimulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of a positional device (PD) (NightBalance, Philips) compared to continuous positive airway pressure (CPAP) in the treatment of OSA assessed by the intergroup differences in apnea hypopnea index (AHI) measured by respiratory polygraphy (RP) | 6 months
  To evaluate the effectiveness of a positional device (PD) (NightBalance, Philips) compared to continuous positive airway pressure (CPAP) in the treatment of OSA by assessing the apnea hypopnea index (AHI) measured by respiratory polygraphy (RP) after 6 months of treatment in a non-inferiority analysis.

SECONDARY OUTCOMES:
Cost-effectiveness of PD in the treatment of OSA compared to CPAP and assessed by the difference in cost between both devices taking into account the AIH measured by RP. | 6 months
  To assess the cost-effectiveness of NightBalance PD in the treatment of OSA compared to CPAP treatment after 6 months of treatment and assessed by the difference in cost between the two treatment methods divided by the difference in effectiveness between the two treatment methods taking into account: AIH (measured by RP)
Cost-effectiveness of PD in the treatment of OSA compared to CPAP and assessed by the difference in cost between both devices taking into account the degree of daytime sleepiness measured by the Epworth scale. | 6 months
  To assess the cost-effectiveness of NightBalance PD in the treatment of OSA compared to CPAP treatment after 6 months of treatment and assessed by the difference in cost between the two treatment methods divided by the difference in effectiveness between the two treatment methods taking into account the degree of daytime sleepiness, measured by the Epworth scale (0-24, where higher scores mean a worse outcome)
Cost-effectiveness of PD in the treatment of OSA compared to CPAP and assessed by the difference in cost between both devices taking into account the quality-adjusted life years measured by the EuroQol-5D questionnaire | 6 months
  To assess the cost-effectiveness of NightBalance PD in the treatment of OSA compared to CPAP treatment after 6 months of treatment and assessed by the difference in cost between the two treatment methods divided by the difference in effectiveness between the two treatment methods taking into account the quality-adjusted life years, measured by the European Quality of Life 5 dimensions (EuroQol-5D) questionnaire (5 dimensions from 1 to 3 points in each one, where higher scores mean a worse outcome)
Cost-effectiveness of PD in the treatment of OSA compared to CPAP and assessed by the difference in cost between both devices taking into account health resources consumed. | 6 months
  To assess the cost-effectiveness of NightBalance PD in the treatment of OSA compared to CPAP treatment after 6 months of treatment and assessed by the difference in cost between the two treatment methods divided by the difference in effectiveness between the two treatment methods taking into account health resources consumed in euros: Initial cost of the device, maintenance costs (consumables, revisions), hospital costs (hospital visits for training, troubleshooting, pressure titration, parameter adjustment, follow-up visits), patient costs (device, consumables, travel).
Conditioned response of PD assesed by the apnea hypopnea index (AHI) measured by respiratory polygraphy (RP) after 1 week and 1 month of withdrawing active treatment | 1 month
  Apnea hypopnea index (AHI) measured by respiratory polygraphy (RP) after 1 week and 1 month of withdrawing active treatment will be assesed and compared to AHI after active treatment with NightBalance for 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cano-Pumarega, MD, PhD, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Pneumology Department, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No